CLINICAL TRIAL: NCT06417255
Title: Comparison Of The Effects Of Kinesiotape Application And Foam Roller Exercises in Individuals With Chronic Low Back Pain
Brief Title: Comparison Of The Effects Of Kinesiotape Application And Foam Roller Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHRONIC LOW BACK PAIN
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotape application (Experimental)
  Interventions: Other: kinesiotape application
- foam roller application (Active Comparator)
  Interventions: Other: foam roller application

INTERVENTIONS:
Other: kinesiotape application — The strips used for kinesiological taping can be applied by giving different shapes. These shapes are I, Y, X, ring (donut), rake and net
  Arms: kinesiotape application
Other: foam roller application — In the foam roller group, "Actifoam" brand non-serrated foam rollers with a size of "15x90" cm were used.
  Arms: foam roller application

SUMMARY:
Low back pain is an important health problem that is common worldwide, with a lifetime prevalence of up to 80%.

DETAILED DESCRIPTION:
Low back pain that lasts less than 6 weeks is called acute low back pain, if it continues for 6-12 weeks it is called subacute low back pain, and if it continues for more than 12 weeks it is called chronic low back pain. The majority of low back pain (97%) is of mechanical origin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic low back pain
* Individuals aged 18-60 years
* Patients without verbal communication barriers
* Patients without cognitive impairment (delirium, dementia, amnesia)

Exclusion Criteria:

* Exercise contraindication (uncontrolled medical conditions)
* Patients with previous spinal surgery
* Patients who develop an allergic reaction to the kinesiotape tape to be applied

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-11 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Measurement with Algometer | 6 weeks
  The algometer, an effective way of measuring pressure pain threshold (PPT), is used to measure soft tissue pain associated with trigger points.
  Pittsburgh Sleep Quality Scale The Pittsburgh Sleep Quality Index is the most commonly used general measure in clinical and research settings to assess sleep quality and quantity. The Pittsburgh Sleep Quality Index (PSQI) consists of a total of 19 questions and 7 components to assess sleep quality during the last month. The total score had a value between 0-21
  Schober Flexibility Test With the patient standing, the examiner marks the spinous process of the first sacral vertebra and 10 cm above this point. The patient is then asked to flex forwards as if trying to touch their toes while keeping their knees straight. If the distance between the two points does not increase by at least 5 cm, this is considered a sign of restriction in lumbar flexion.
Pittsburgh Sleep Quality Scale | 6 weeks
  The Pittsburgh Sleep Quality Index is the most commonly used general measure in clinical and research settings to assess sleep quality and quantity. The Pittsburgh Sleep Quality Index (PSQI) consists of a total of 19 questions and 7 components to assess sleep quality during the last month. The total score had a value between 0-21
Schober Flexibility Test | 6 weeks
  With the patient standing, the examiner marks the spinous process of the first sacral vertebra and 10 cm above this point. The patient is then asked to flex forwards as if trying to touch their toes while keeping their knees straight. If the distance between the two points does not increase by at least 5 cm, this is considered a sign of restriction in lumbar flexion.
The finger-to-floor distance | 6 weeks
  The finger-to-floor distance test is a test that measures specific physical disability. This test is performed with the person standing upright with feet together. The patient is asked to lean as far forward as possible with knees, arms and fingers fully extended. The vertical distance between the tip of the middle finger and the floor is measured with a flexible tape measure.
Tampa Kinesiophobia Fatigue Scale | 6 weeks
  The Tampa Kinesiophobia Scale measures fear of movement and fear of (re)injury during movement. High fear of movement and/or (re)injury, as measured by the Tampa Kinesiophobia Scale, has been found to be associated with poor performance on a number of physical tests.
  The minimum and maximum values of the Tampa Kinesiophobia Fatigue Scale are between 17 and 68. The total score range of this scale is between 0 and 68.
Oswestry Scale | 6 weeks
  The Oswestry Disability Index, first introduced by Fairbank et al. in 1980, is considered close to the gold standard for measuring the severity of disability due to low back pain. The Oswestry scale is a self-administered, free, easy-to-use and easy-to-score questionnaire containing 10 questions on different functional domains.
  The Oswestry Disability Index (ODI) is a widely used tool to assess disability related to low back pain. It consists of 10 sections addressing various daily activities, each scored on a scale of 0 to 5. The minimum score is 0, indicating no disability, while the maximum score is 50, indicating severe disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hazal GENÇ, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No